CLINICAL TRIAL: NCT05480540
Title: The Effect of Serious Game-Based and Video-Assisted Practices in Sterile Dressing and Surgical Instrument Preparation Education on Nursing Students' Knowledge, Skills and Anxiety Levels
Brief Title: The Effect of Serious Games
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Cemile AKTUG, Head of Otolaryngology, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-95674917-108.99-92819
Record Dates: First submitted 2022-07-21; First posted 2022-07-29 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Operating Room Nursing; Serious Game; Education; Surgical Instrument; Sterile Dressing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious game (Experimental): A serious game-based web application on Sterile Dressing and Surgical Instrument Preparation Training, which was prepared in accordance with the formal education curriculum and prepared as a support for formal education, will be downloaded to the mobile phones of the students in the intervention group.
  Interventions: Behavioral: Serious game
- Video (Active Comparator): The video prepared on sterile dressing and surgical instrument preparation training will be shown to the students in the control group for 2 weeks.
  Interventions: Behavioral: Serious game

INTERVENTIONS:
Behavioral: Serious game — According to the curriculum, as of the third week, a serious game-based web application on Sterile Dressing and Surgical Instrument Preparation Training, which is prepared in accordance with the formal education curriculum and prepared as a support for formal education, will be downloaded to the mobile phones of the students in the intervention group as of the third week. Students would be informed that they could use the application for two weeks whenever they wanted and as much as they wanted.

SUMMARY:
Today, there is a need to integrate and restructure rapidly developing technology into teaching environments. When web-based applications, which are among the popular and innovative technologies, are examined, it is seen that they are used in many areas of education. In this study, it was aimed to evaluate the effects of sterile hand washing, sterile dressing, sterile package opening and surgical instrument preparation training on anxiety, satisfaction, knowledge and skill levels by designing a serious game-based web application that allows nursing students to gain skills and practice in psychomotor applications. The universe of the study will consist of students enrolled in the Operating Room Nursing course in the Nursing Department of the Faculty of Health Sciences of Gümüşhane University in the spring semester of the 2021-2022 academic year, and the sample will consist of 94 students who meet the study criteria and agree to participate in the study. Data; It will be collected with the Introductory Characteristics Form, Operating Room Applications Information Form, Sterile Dressing and Surgical Instrument Preparation Skills Checklist, State Trait Anxiety Scale (WHO) and Visual Comparison Scale (GLO). Oral lectures will be given to all students by the instructor in charge of the course for two hours a week for two weeks, according to the lesson plan. Before the oral presentation, the 'Student Information Form' and the 'Operating Room Applications Information Form' will be applied to the students. After the questionnaire applications, the students will be divided into two groups, 47 students in the intervention group and 47 students in the control group, by randomization method. A serious game-based web application will be downloaded to the mobile phones of the students in the intervention group, on sterile dressing and surgical instrument preparation training, prepared in accordance with the formal education curriculum. How to use it will be shown. The students in the control group will be shown the video prepared by the researcher on sterile dressing and surgical instrument preparation training. Students in both groups will be informed that they can use this application for two weeks whenever they want and as much as they want. At the end of two weeks, a skill test will be given to the control and intervention groups in the laboratory. WHO will be applied to both groups before and after the skill test. Immediately after the skill test, the Operating Room Applications Information Form will be applied to both groups to measure the level of knowledge, the State Anxiety Inventory (DBS) to determine their anxiety level, and the GAS to measure satisfaction. Three weeks after the first skill test, students' second skill measures will be evaluated using the 'Surgical Instrument Preparation Skill Checklist', and their anxiety levels will be evaluated with the Trait Anxiety Inventory. The obtained data will be analyzed with appropriate statistical methods using the SPSS for Windows 23.0 program (Statistical Package for the Social Sciences)

ELIGIBILITY:
Inclusion Criteria:

* Registering for the first time HEMSEC218 Operating Room Nursing course,
* Having internet access,
* Volunteering to participate in the study,
* Smart phone, computer or tablet etc. that can activate the game. have one of the tools

Exclusion Criteria:

* To have received training (in-service training, courses, seminars, etc.) related to operating room nursing,
* Having graduated from a health vocational high school and having experience in the operating room,
* Taking the HEMSEC218 Operating Room Nursing course for the second time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Outcome 1 | 12 months
  Sterile Dressing and Surgical Instrument Preparation at knowledge level

SECONDARY OUTCOMES:
Outcome 2 | 12 months
  Sterile Dressing and Surgical Instrument Preparation skill level